CLINICAL TRIAL: NCT05064865
Title: Impact of Regular Consumption of Grapes on Eye Health in Singapore Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S15
Record Dates: First submitted 2021-08-30; First posted 2021-10-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Eye Health; Age-related Macular Degeneration
Keywords: Eye Health; Age-related Macular Degeneration; carotenoids
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-dried table grape powder (Experimental): The intervention group will consume 46 g/day of a freeze-dried table grape powder.
  Interventions: Dietary Supplement: Freeze-dried table grape powder
- Placebo grape powder (Placebo Comparator): The control group will consume the same amount of a placebo with a similar taste to the table grape powder.
  Interventions: Dietary Supplement: Placebo of the table grape powder

INTERVENTIONS:
Dietary Supplement: Freeze-dried table grape powder — Consumption of 46g/day freeze-dried table grape powder
  Arms: Freeze-dried table grape powder
Dietary Supplement: Placebo of the table grape powder — Consumption of 46g/day placebo version of the freeze-dried table grape powder
  Arms: Placebo grape powder

SUMMARY:
Aging epidemics in Singapore are rapidly increasing and Age-related macular degeneration (AMD) prevalence is significantly associated with older age. This study aims to understand the effect of consuming freeze-dried table grape powder on AMD in an older population.

DETAILED DESCRIPTION:
This will be carried out through a 16-week double-blind, randomized, placebo-controlled trial of parallel study design. Thirty-eight men and women (aged between 60 and 85 years old inclusive) will recruited and assigned to an intervention or placebo group. The intervention group will consume 46 g/day of a freeze-dried table grape and the control group will consume the same amount of a placebo, table grape placebo powder. Measurements of 1) macular pigment optical density (MPOD), a clinical marker for eye health, 2) carotenoids status, 3) markers of oxidative stress, 4) markers of endothelial function, 5) body size and blood pressure, and 6) dietary assessment will be assessed over the 16-week study. This study will consist of 1 screening visit and 5 study visits in 4-week intervals to the Food Science and Technology Department, Occupational Health Clinic and National University Heart Centre.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, aged between 60 and 85 years old inclusive
* Able to give informed consent in English

Exclusion Criteria:

* Smokers
* Allergy to grapes
* Known eye diseases (macular degeneration, cataracts, retinopathy or glaucoma), blindness in at least one eye or have had eye surgery
* Abnormal kidney and liver function
* Taking eye medication and/or dietary supplements for the eyes for the past 3 months
* Taking supplements containing carotenoids (e.g. Vitamin A, lutein, zeaxanthin) for the past 3 months
* Currently on type 2 diabetic medication.
* Currently on anti-hypertensive or cholesterol-lowering; unless this prescription has been ongoing for more than 3 years prior to study participation.
* Currently on a specialized diet (e.g. vegetarian, vegan, weight loss diet, low fat diet)
* Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine, 340ml of beer/cider or 45ml of distilled spirit.
* Significant change in weight (≥ 3 kg body weight) in the past 3 months
* Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week
* Poor peripheral venous access based on past experiences with blood draw
* Participating in another clinical study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in macular pigment optical density | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Macular pigment optical density will be measured using macular pigment scanner
Change in skin carotenoid status | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Skin carotenoid status (a.u) measured using NuSkin II, resonance Raman spectroscopy
Change in blood carotenoid concentration | Every eight weeks (week 0, week 8, week 16)
  Blood carotenoid concentration to be quantified by HPLC

SECONDARY OUTCOMES:
Change in flow mediate dilation | week 0 and week 16
  Flow mediate dilation (%)
Change in endothelial function | week 0 and week 16
  Endothelial functions are determined by the function of endothelial progenitor cells
Change in the concentration if Endothelin-1 in plasma | week 0 and week 16
  Endothelin-1 concentration
Change in the concentration if Nitric Oxide in plasma | week 0 and week 16
  Nitric Oxide concentration
Change in body weight | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Body weight (kg) measured using body scale
Change in BMI | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Weight and height will be combined to report BMI in kg/m^2
Change in blood pressure | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Systolic and diastolic blood pressure (mmHg) measured using sphygmomanometer
change in waist circumference | Every four weeks (week 0, week 4, week 8, week 12, week 16)
  Waist circumference (cm) measured using measuring tape
Change in the concentration of malondialdehyde in plasma | Every eight weeks (week 0, week 8, week 16)
  Malondialdehyde concentration
Change in the concentration of 8-iso-prostaglandin F2α in plasma | Every eight weeks (week 0, week 8, week 16)
  8-iso-prostaglandin F2α concentration
Change in blood glucose concentration | Every eight weeks (week 0, week 8, week 16)
  Blood glucose concentration (mmol/l)
Change in total cholesterol | Every eight weeks (week 0, week 8, week 16)
  Total cholesterol (mmol/l)
Change in high-density lipoprotein cholesterol | Every eight weeks (week 0, week 8, week 16)
  High-density lipoprotein cholesterol (mmol/l)
Change in low-density lipoprotein cholesterol | Every eight weeks (week 0, week 8, week 16)
  Low-density lipoprotein cholesterol (mmol/l)
Change in total triglyceride | Every eight weeks (week 0, week 8, week 16)
  Total triglyceride (mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be key data will be de-identified prior to statistical analysis

REFERENCES:
- [Background] Gehrs KM, Anderson DH, Johnson LV, Hageman GS. Age-related macular degeneration--emerging pathogenetic and therapeutic concepts. Ann Med. 2006;38(7):450-71. doi: 10.1080/07853890600946724. PMID 17101537
- [Derived] Hu W, Zheng R, Feng Y, Tan D, Chan Chung-Tsing G, Su X, Kim JE. Impacts of regular consumption of grapes on macular pigment accumulation in Singapore older adults: a randomized controlled trial. Food Funct. 2023 Sep 19;14(18):8321-8330. doi: 10.1039/d3fo02105j. PMID 37605542